CLINICAL TRIAL: NCT04878432
Title: Single-arm, Open Label, Phase II Study of MBG453 (Sabatolimab) Added to FDA Approved Hypomethylating Agents of Investigator's Choice (IV/SC/Oral) for Patients With Intermediate, High or Very High Risk Myelodysplastic Syndrome (MDS) as Per IPSS-R Criteria (US Multi-center) (STIMULUS MDS-US)
Brief Title: STIMULUS MDS-US : Sabatolimab Added to HMA in Higher Risk MDS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of efficacy in the program as demonstrated in the earlier CMBG453B12301 (STIMULUS MDS-2) study.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMBG453B1US01
Record Dates: First submitted 2021-05-05; First posted 2021-05-07 (Actual); Results first posted 2025-07-31 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Myelodysplastic Syndrome (MDS)
Keywords: sabatolimab; phase II; MBG453; TIM-3; decitabine; azacitidine; oral decitabine; INQOVI; myelodysplastic syndrome (MDS); adult; MDS
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — sabatolimab; Azacitidine; Decitabine; decitabine and cedazuridine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MBG453 (sabatolimab) + HMA (Experimental): MBG453 (sabatolimab) + HMA of investigator's choice (IV Decitabine or Azacitidine /SC Azacitidine /Oral Decitabine (cedazuridine combination (INQOVI)))
  Interventions: Drug: MBG453; Drug: Azacitidine; Drug: Decitabine; Drug: INQOVI (oral decitabine)

INTERVENTIONS:
Drug: MBG453 — Solution for intravenous infusion
  Other Names: sabatolimab
Drug: Azacitidine — Solution for subcutaneous injection or intravenous administration
Drug: Decitabine — Solution for intravenous administration
Drug: INQOVI (oral decitabine) — Tablet for oral administration

SUMMARY:
The main objective of this study was to assess the safety profile of MBG453 (sabatolimab) in combination with FDA approved hypomethylating agents (HMAs) of investigator's choice (IV Decitabine or Azacitidine /SC Azacitidine /Oral Decitabine (cedazuridine combination (INQOVI))).

DETAILED DESCRIPTION:
This was a single arm, nonrandomized, open label, Phase II multicenter study of i.v sabatolimab added to FDA approved HMA agents of Investigator's choice (i.v/s.c/oral) in adult patients with intermediate, high or very high risk MDS as per IPSS-R criteria.

There were 4 separate periods of this study:

1. Screening period (signing of written informed consent through day of enrollment),
2. Core phase for up to 12 months,
3. Extension phase for efficacy and/or survival status (up to 12 months after the core phase),
4. Post-treatment safety follow-up period monitoring for AEs for 30 days following the last dose of azacitidine or decitabine or INQOVI (oral decitabine), or 150 days following the last dose of sabatolimab, whichever was later.

During the conduct of the study there were 2 updates to the Novartis development strategy for sabatolimab. Based on the results from the Phase II STIMULUS MDS-1 study, recruitment was halted for CMBG453B1US01 (STIMULUS MDS-US) on 30-Sep-2022. Novartis confirmed the decision to halt recruitment was not based on any safety findings or safety concerns. Patients who were on study treatment or in follow-up were continued as per the protocol. Furthermore, on 11-Jan-2024, all sabatolimab investigators were notified by Novartis that, based on decision taken in Dec-2023, that the sabatolimab development program (which included study CMBG453B1US01) would be terminated. After the decision was made to discontinue the sabatolimab development program, participants already enrolled in the CMBG453B1US01 study were prepared for closure; these close out activities took approximately 9 months. The actual last patient last visit date was 1 Sep 2024.

ELIGIBILITY:
Key inclusion criteria:

1. Signed informed consent was obtained prior to participation in the study.
2. Age ≥ 18 years at the date of signing the informed consent form (ICF).
3. Morphologically confirmed diagnosis of a myelodysplastic syndrome (MDS) primary or secondary based on 2016 WHO classification by Investigator assessment with one of the following prognostic risk categories, based on the International Prognostic Scoring System (IPSS-R).. Note: MDS diagnosis history were recorded in the CRF:

   * Very high (> 6 points)
   * High (> 4.5 to ≤ 6 points)
   * Intermediate (> 3 to ≤ 4.5 points)
4. Not suitable at the time of Screening for immediate myeloablative/chemotherapy or HSCT based on Investigator assessment of age, comorbidities, local guidelines, institutional practice (any or all of these).
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2.
6. AST and ALT ≤ 3 × upper limit of normal (ULN).
7. Total bilirubin ≤ 2 × ULN (except in the setting of isolated Gilbert syndrome).
8. Estimated glomerular filtration rate ≥ 30 mL/min/1.73 m2 (estimation based on modification of diet in renal disease formula, by local laboratory).
9. Patient was able to communicate with the Investigator and had the ability to comply with the requirements of the study procedures.

Key exclusion criteria

1. Prior exposure to TIM-3 directed therapy at any time. Prior therapy with immune checkpoint inhibitors (e.g., anti-CTLA4, anti-PD-1, anti-PD-L1, or anti-PD-L2), cancer vaccines were allowed only if the last dose of the drug was administered more than 4 months prior to enrollment.
2. Previous treatment for intermediate, high or very high risk MDS (based on IPSS-R) with chemotherapy or other antineoplastic agents including lenalidomide and hypomethylating agent (HMAs) such as decitabine or INQOVI (oral decitabine) or azacitidine (patients who had up to 1 cycle of HMAs were included). However, previous treatment with hydroxyurea was permitted.
3. Diagnosis of acute myeloid leukemia (AML) including acute promyelocytic leukemia and extra-medullary acute myeloid leukemia based on WHO 2016 classification.
4. Diagnosis of Chronic myelomonocytic leukemia (CMML), or primary or secondary myelofibrosis based on 2016 WHO classification.
5. History of organ transplant or allogenic HSCT.
6. Patients with prior malignancy, except:

   1. Patients with history of lower risk Myelodysplastic syndrome (MDS) treated by supportive care (e.g., growth factors, transforming growth factor- beta agents) or untreated were eligible.
   2. Patients with history of lower risk MDS who were treated adequately with lenalidomide and then failed were eligible.
   3. Patients with history of adequately treated malignancy for which no anticancer systemic therapy (namely chemotherapy, radiotherapy or surgery) was ongoing or required during the course of the study. Patients who were receiving adjuvant therapy such as hormone therapy were eligible.
7. Patients with MDS based on 2016 WHO classification with revised International Prognostic Scoring System (IPSS-R) ≤ 3.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2022-03-17 (Actual); Primary Completion 2023-10-26 (Actual); Study Completion 2024-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (15):
- United States (15):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Arizona Oncology Associates, Tucson, Arizona
  - SCRI-Colorado Blood Cancer Institute, Denver, Colorado
  - Yale University School Of Medicine, New Haven, Connecticut
  - Advent Health Orlando, Orlando, Florida
  - Uni of Massachusetts Medical Center, Worcester, Massachusetts
  - University Of Michigan, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - Tisch Hospital NYU Langone, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Duke Cancer Institute, Durham, North Carolina
  - University Hospitals Of Cleveland, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Uni Of TX MD Anderson Cancer Cntr, Houston, Texas
  - Texas Oncology San Antonio USO, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on https://www.clinicalstudydatarequest.com/.
URL: https://www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2688

RESULTS

PARTICIPANT FLOW:
Groups:
- MBG453 (Sabatolimab) + Hypomethylating Agents (HMA): MBG453 400 mg/4 ml + HMA (azacitidine 75 mg/m^2, decitabine 20 mg/m^2, or INQOVI (oral decitabine) 100 mg cedazuridine/35 mg)
Period: Overall Study
Arm/Group | MBG453 (Sabatolimab) + Hypomethylating Agents (HMA)
Started | 39
Completed | 2
Not Completed | 37
Not completed — Adverse Event | 1
Not completed — Death | 2
Not completed — Unsatisfactory Therapeutic Effect | 3
Not completed — Withdrawal by Subject | 6
Not completed — Progressive Disease | 7
Not completed — New Therapy for Study Indication | 7
Not completed — Physician Decision | 11

BASELINE CHARACTERISTICS:
Arm/Group | MBG453 (Sabatolimab) + Hypomethylating Agents (HMA)
Number analyzed (Participants) | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 25
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.8 (11.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 31
  More than one race | 0
  Unknown or Not Reported | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events and Serious Adverse Events
Description: An adverse event (AE) is any untoward medical occurrence (e.g. any unfavorable and unintended sign [including abnormal laboratory findings], symptom or disease) in a participant or clinical investigation participant after providing written informed consent for participation in the study. Therefore, an AE may or may not be temporally or causally associated with the use of a medicinal (investigational) product.
Time Frame: Adverse events are reported from the first dose of study medication up to approximately 24 months plus 30 - 150 day safety follow up dependent on HMA, for a maximum timeframe of approximately 29 months.
Population: Safety set - The SS included all patients who received at least one dose of any component of the study medication (sabatolimab+HMA).
Measure: Count of Participants; unit: Participants
Arm/Group | MBG453 (Sabatolimab) + Hypomethylating Agents (HMA)
Number analyzed (Participants) | 39
Participants
  Adverse events (AEs) | 39
  Treatment-related Adverse events | 30
  AEs with grade ≥ 3 | 35
  Treatment-related AEs with grade ≥ 3 | 25
  Serious Adverse Events (SAEs) | 23
  Treatment-related SAEs | 8
  Fatal SAEs | 0
  Treatment-related Fatal SAEs | 0
  AEs leading to discontinuation | 3
  Treatment-related AEs leading to discontinuation | 3
  AEs leading to dose adjustment/interruption | 8
  AEs requiring additional therapy | 32

2. Secondary Outcome: Number of Participants With Complete Remission According to International Working Group (IWG) for MDS (2006) With MBG453 (Sabatolimab) in Combination With HMAs (IV/SC/Oral) by 12 Months.
Description: Complete remission rate was assessed according to International Working Group (IWG) for MDS (2006) with MBG453 (sabatolimab) in combination with HMAs (IV/SC/Oral) in Participants with intermediate, high, or very high risk MDS by 12 months.
Time Frame: up to Month 12
Population: Full analysis set - The FAS comprised all enrolled patients who received any component of the study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | MBG453 (Sabatolimab) + Hypomethylating Agents (HMA)
Number analyzed (Participants) | 39
Participants | 1

3. Secondary Outcome: Number of Participants With Progression Free Survival - Death and Disease Progression
Description: Defined as time from enrollment to disease progression (including transformation to leukemia per WHO 2016 classification), relapse from CR according to IWG-MDS or death due to any cause, whichever occurs first, as per investigator assessment by 12 months post last patient first treatment (LPFT).
Time Frame: up to Month 24
Population: Full analysis set - The FAS comprised all enrolled patients who received any component of the study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | MBG453 (Sabatolimab) + Hypomethylating Agents (HMA)
Number analyzed (Participants) | 39
Participants
  Death | 7
  Disease Progression | 9

4. Secondary Outcome: Progression Free Survival - 50th Percentile
Description: as for outcome 3
Time Frame: up to Month 24
Population: Full analysis set - The FAS comprised all enrolled patients who received any component of the study medication.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | MBG453 (Sabatolimab) + Hypomethylating Agents (HMA)
Number analyzed (Participants) | 39
months | 11.56 [4.24 to 16.59]

5. Secondary Outcome: Progression Free Survival - Percent Probability - Kaplan-Meier Probability Estimates
Description: as for outcome 3
Time Frame: Months 6 and 12
Population: Full analysis set - The FAS comprised all enrolled patients who received any component of the study medication.
Measure: Number (95% Confidence Interval); unit: percent probability
Arm/Group | MBG453 (Sabatolimab) + Hypomethylating Agents (HMA)
Number analyzed (Participants) | 39
percent probability
  6 months | 65.28 [43.18 to 80.53]
  12 months | 43.27 [19.45 to 65.14]

6. Secondary Outcome: Overall Survival - Number of Participants Who Died
Description: Overall Survival (OS) is defined as the time from the first dose of study medication to death due to any cause.
Time Frame: up to Month 24
Population: Full analysis set - The FAS comprised all enrolled patients who received any component of the study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | MBG453 (Sabatolimab) + Hypomethylating Agents (HMA)
Number analyzed (Participants) | 39
Participants | 20

7. Secondary Outcome: Overall Survival - 50th Percentile
Description: Overall Survival (OS) is defined as the time from the first dose of study medication to death due to any cause.
Time Frame: up to Month 24
Population: Full analysis set - The FAS comprised all enrolled patients who received any component of the study medication.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | MBG453 (Sabatolimab) + Hypomethylating Agents (HMA)
Number analyzed (Participants) | 39
months | 15.77 [8.74 to 19.19]

8. Secondary Outcome: Overall Survival - Percent Probability - Kaplan-Meier Probability Estimates
Description: Overall Survival (OS) is defined as the time from the first dose of study medication to death due to any cause.
Time Frame: up to Month 24
Population: Full analysis set - The FAS comprised all enrolled patients who received any component of the study medication.
Measure: Number (95% Confidence Interval); unit: percent probability
Arm/Group | MBG453 (Sabatolimab) + Hypomethylating Agents (HMA)
Number analyzed (Participants) | 39
percent probability
  6 months | 82.90 [65.77 to 91.95]
  9 months | 65.66 [46.24 to 79.50]
  12 months | 61.56 [41.79 to 76.35]
  15 months | 53.35 [33.57 to 69.65]
  18 months | 35.57 [16.40 to 55.37]
  21 months | 28.45 [10.67 to 49.37]
  24 months | 21.34 [6.07 to 42.68]

9. Secondary Outcome: Leukemia-free Survival - Number of Participants Who Died and Number of Participants Who Progressed to Leukemia
Description: Leukemia-free survival (LFS) is the time from the date of the first dose of medication to ≥ 20% blasts in bone marrow/peripheral blood (per WHO 2016 classification) or death due to any cause.
Time Frame: up to Month 24
Population: Full analysis set - The FAS comprised all enrolled patients who received any component of the study medication.
Measure: Number; unit: Participants
Arm/Group | MBG453 (Sabatolimab) + Hypomethylating Agents (HMA)
Number analyzed (Participants) | 39
Participants
  Death | 16
  Progressed to leukemia | 6

10. Secondary Outcome: Leukemia-free Survival - 50th Percentile
Description: as for outcome 9
Time Frame: up to Month 24
Population: Full analysis set - The FAS comprised all enrolled patients who received any component of the study medication.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | MBG453 (Sabatolimab) + Hypomethylating Agents (HMA)
Number analyzed (Participants) | 39
months | 11.30 [6.01 to 16.59]

11. Secondary Outcome: Leukemia-free Survival - Percent Probability - Kaplan-Meier Probability Estimates
Description: as for outcome 9
Time Frame: Months 6 and 12
Population: Full analysis set - The FAS comprised all enrolled patients who received any component of the study medication.
Measure: Number (95% Confidence Interval); unit: percent probability
Arm/Group | MBG453 (Sabatolimab) + Hypomethylating Agents (HMA)
Number analyzed (Participants) | 39
percent probability
  6 months | 70.58 [50.67 to 83.65]
  12 months | 48.04 [27.46 to 65.98]

12. Secondary Outcome: Percentage of Participants With Complete Remission, Marrow Complete Remission and/or Partial Remission
Description: Percentage of complete remission, marrow complete remission, and/or partial remission according to IWG-MDS remission criteria as per investigator assessment
Time Frame: up to Month 24
Population: Full analysis set - The FAS comprised all enrolled patients who received any component of the study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | MBG453 (Sabatolimab) + Hypomethylating Agents (HMA)
Number analyzed (Participants) | 39
Participants
  Complete Remission (CR) | 1
  Marrow Complete Remission (mCR) | 6
  mCR with hematological improvement (HI) | 4
  Partial Remission (PR) | 2
  Stable Disease (SD) | 11
  SD with hematological improvement (HI) | 1
  CR+mCR+PR | 9
  CR+PR+HI | 8
  CR+mCR+PR+HI | 10

13. Secondary Outcome: Time to Complete Remission
Description: Time to Complete Remission is defined as the time from the date of the first dose of study medication to the first documented CR.
Time Frame: up to Month 24
Population: Full analysis set - The FAS comprised all enrolled patients who received any component of the study medication and who had complete remission.
Measure: Median (Standard Deviation); unit: months
Arm/Group | MBG453 (Sabatolimab) + Hypomethylating Agents (HMA)
Number analyzed (Participants) | 1
months | 5.91 (NA) — Not applicable for a single patient who met this condition.

14. Secondary Outcome: Improvement in Packed RBCs Transfusion Independence - Mean Total Duration (Weeks) of Transfusion Independence Post-baseline
Description: RBC/Platelets transfusion independence is defined as a participant having received <0 units RBC/Platelets transfusions during at least 8 consecutive weeks after enrollment.
Time Frame: up to Month 24
Population: Full analysis set - The FAS comprised all enrolled patients who received any component of the study medication.
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | MBG453 (Sabatolimab) + Hypomethylating Agents (HMA)
Number analyzed (Participants) | 39
weeks | 27.02 (21.194)

15. Secondary Outcome: Number of Participants With Improvement in Packed RBCs Transfusion Independence - At Least One Period of Transfusion Independence Post Baseline
Description: RBC/Platelets transfusion independence rate is defined as the percentage of participants having received <0 units RBC/Platelets transfusions during at least 8 consecutive weeks after enrollment.
Time Frame: up to Month 24
Population: Full analysis set - The FAS comprised all enrolled patients who received any component of the study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | MBG453 (Sabatolimab) + Hypomethylating Agents (HMA)
Number analyzed (Participants) | 39
Participants | 25

16. Secondary Outcome: Improvement in Platelets Transfusion Independence - Mean Total Duration (Weeks) of Transfusion Independence Post-baseline
Description: as for outcome 14
Time Frame: up to Month 24
Population: Full analysis set - The FAS comprised all enrolled patients who received any component of the study medication.
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | MBG453 (Sabatolimab) + Hypomethylating Agents (HMA)
Number analyzed (Participants) | 39
weeks | 27.41 (22.397)

17. Secondary Outcome: Number of Participants With Improvement in Platelets Transfusion Independence - At Least One Period of Transfusion Independence Post Baseline
Description: RBC/Platelets transfusion independence rate is defined as the proportion of participants having received <0 units RBC/Platelets transfusions during at least 8 consecutive weeks after enrollment.
Time Frame: up to Month 24
Population: Full analysis set - The FAS comprised all enrolled patients who received any component of the study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | MBG453 (Sabatolimab) + Hypomethylating Agents (HMA)
Number analyzed (Participants) | 39
Participants | 27

18. Post Hoc Outcome: All Collected Deaths
Time Frame: Deaths are reported from the first dose of study medication up to approximately 24 months plus 30 - 150 day safety follow up dependent on HMA, for a maximum timeframe of approximately 29 months.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | MBG453 (Sabatolimab) + Hypomethylating Agents (HMA)
Number analyzed (Participants) | 39
Participants
  On-treatment Deaths | 2
  Off-treatment Deaths | 18
  Total Deaths | 20

ADVERSE EVENTS:
Time Frame: Adverse events are reported from the first dose of study medication up to approximately 24 months plus 30 - 150 day safety follow up dependent on HMA, for a maximum timeframe of approximately 29 months.
Description: This was a single arm study. The study drugs of the hypomethylating agents decitabine, azacitidine, and oral decitabine (cedazuridine/decitabine) were considered to be clinically equivalent towards the standard of care for the treatment of higher risk Myelodysplastic syndrome at the doses administered; therefore, these were reported in the same arm. The study had a small sample size and was not powered to separate into different arms by design.
Groups:
- MBG453+HMA: MBG453 400 mg/4 ml + HMA (azacitidine 75 mg/m^2, decitabine 20 mg/m^2, or INQOVI (oral decitabine) 100 mg cedazuridine/35 mg)
Arm/Group | MBG453+HMA
All-Cause Mortality (participants affected / at risk) | 20/39
Serious Adverse Events (participants affected / at risk) | 23/39
Other Adverse Events (participants affected / at risk) | 35/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MBG453+HMA (N=39)
Febrile neutropenia (Blood and lymphatic system disorders) | 14
Immune thrombocytopenia (Blood and lymphatic system disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 2
Sinus tachycardia (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Photopsia (Eye disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2
Haematochezia (Gastrointestinal disorders) | 1
Proctitis (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Malaise (General disorders) | 1
Physical deconditioning (General disorders) | 1
Pyrexia (General disorders) | 2
Bacteraemia (Infections and infestations) | 1
COVID-19 (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Device related infection (Infections and infestations) | 1
Enterocolitis infectious (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 5
Sepsis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 2
Fall (Injury, poisoning and procedural complications) | 2
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Hypervolaemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Encephalopathy (Nervous system disorders) | 1
Delirium (Psychiatric disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Penile ulceration (Skin and subcutaneous tissue disorders) | 1
Embolism (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MBG453+HMA (N=39)
Anaemia (Blood and lymphatic system disorders) | 16
Febrile neutropenia (Blood and lymphatic system disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 4
Anorectal discomfort (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 15
Diarrhoea (Gastrointestinal disorders) | 8
Dry mouth (Gastrointestinal disorders) | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 11
Stomatitis (Gastrointestinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 3
Chills (General disorders) | 6
Fatigue (General disorders) | 12
Oedema peripheral (General disorders) | 7
Pyrexia (General disorders) | 5
Sinusitis (Infections and infestations) | 2
Tooth infection (Infections and infestations) | 2
Contusion (Injury, poisoning and procedural complications) | 4
Fall (Injury, poisoning and procedural complications) | 6
Infusion related reaction (Injury, poisoning and procedural complications) | 4
Skin abrasion (Injury, poisoning and procedural complications) | 2
Blood bilirubin increased (Investigations) | 2
Blood creatinine increased (Investigations) | 2
Lipase increased (Investigations) | 2
Lymphocyte count decreased (Investigations) | 3
Neutrophil count decreased (Investigations) | 15
Platelet count decreased (Investigations) | 16
Weight decreased (Investigations) | 2
White blood cell count decreased (Investigations) | 16
Abnormal loss of weight (Metabolism and nutrition disorders) | 4
Decreased appetite (Metabolism and nutrition disorders) | 4
Gout (Metabolism and nutrition disorders) | 2
Hyperphosphataemia (Metabolism and nutrition disorders) | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 6
Hypomagnesaemia (Metabolism and nutrition disorders) | 3
Hyponatraemia (Metabolism and nutrition disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Back pain (Musculoskeletal and connective tissue disorders) | 6
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Joint swelling (Musculoskeletal and connective tissue disorders) | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Dizziness (Nervous system disorders) | 7
Dysgeusia (Nervous system disorders) | 4
Headache (Nervous system disorders) | 12
Hypoaesthesia (Nervous system disorders) | 2
Tremor (Nervous system disorders) | 2
Anxiety (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 6
Dysuria (Renal and urinary disorders) | 3
Haematuria (Renal and urinary disorders) | 2
Pollakiuria (Renal and urinary disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 5
Pruritus (Skin and subcutaneous tissue disorders) | 7
Rash (Skin and subcutaneous tissue disorders) | 3
Hot flush (Vascular disorders) | 2
Hypertension (Vascular disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2023-02-08): https://cdn.clinicaltrials.gov/large-docs/32/NCT04878432/Prot_000.pdf
  • Statistical Analysis Plan (2025-02-07): https://cdn.clinicaltrials.gov/large-docs/32/NCT04878432/SAP_001.pdf